CLINICAL TRIAL: NCT04938180
Title: A Phase 2, Adaptive, Open-Label, Multiple-Dose, Dose-Escalation Study to Evaluate the Efficacy, Safety, Tolerability, and Pharmacokinetics of Intravenous AMB-05X in Subjects With Tenosynovial Giant Cell Tumor
Brief Title: A Phase 2 Study of Intravenous AMB-05X in Tenosynovial Giant Cell Tumor Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Further enrollment was halted in November 2021, enrolled subjects completed the study. Sponsor stopped further recruitment in this intravenous study to focus on intra-articular route of administration in subjects with tenosynovial giant cell tumor.
Sponsor: AmMax Bio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMB-051-02
Record Dates: First submitted 2021-06-16; First posted 2021-06-24 (Actual); Results first posted 2024-05-24 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Tenosynovial Giant Cell Tumor; Pigmented Villonodular Synovitis; TGCT; PVNS - Pigmented Villonodular Synovitis
Keywords: Tenosynovial Giant Cell Tumor, TGCT, PVNS
MeSH Terms: conditions — Giant Cell Tumor of Tendon Sheath; Synovitis, Pigmented Villonodular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cohort A (Experimental): Each subject will receive a low dose of AMB-05X every 2 weeks, for a total of 6 doses over the 12-week treatment period.
  Interventions: Biological: AMB-05X

INTERVENTIONS:
Biological: AMB-05X — AMB-05X is a fully human antibody antagonist (immunoglobulin G, type 2 [IgG2]) specific to the extracellular domain of human CSF1R

SUMMARY:
The purpose of this Phase 2, open-label, multiple-dose, dose-escalation study is to evaluate intravenous AMB-05X in the treatment of subjects with TGCT.

DETAILED DESCRIPTION:
AMB-05X drug substance is a human monoclonal antibody against the colony-stimulating factor 1 receptor (CSF1R).

ELIGIBILITY:
Inclusion Criteria:

1. Subject ≥ 18 years
2. A confirmed diagnosis of TGCT
3. Measurable disease based on RECIST v1.1
4. Symptomatic disease
5. Stable prescription of analgesic regimen
6. Agrees to follow contraception guidelines
7. Adequate hematologic, hepatic, and renal function, at Screening
8. Willing and able to complete self-assessment instruments throughout the study

Exclusion Criteria:

1. Prior investigational drug use within 4 weeks or 5 half-lives of Baseline
2. Current or prior radiotherapy within 3 months before Baseline
3. Current or prior active cancer within 3 years before Baseline that requires/required therapy (eg, surgery, chemotherapy, or radiation therapy)
4. Known metastatic TGCT or malignant transformation of diffuse-type TGCT
5. Hepatitis C virus (HCV) or hepatitis B virus (HBV) or known active or chronic infection with human immuno deficiency virus (HIV)
6. Known active tuberculosis (TB)
7. Significant concomitant arthropathy in the affected joint, serious illness, uncontrolled infection, or a medical or psychiatric history
8. Women who are pregnant or breastfeeding
9. Screening Fridericia-corrected QT interval(QTcF) ≥450ms (men) or ≥470ms (women)
10. MRI contraindications (eg, pacemaker, loose metallic implants)
11. History of hypersensitivity to any ingredient in the study drug
12. History of drug or alcohol abuse within 3 months before Baseline
13. Has any other severe acute or chronic medical or psychiatric condition or clinically significant laboratory abnormality that may increase the risk associated with study participation/treatment, interfere with interpretation of study results, or, in the Investigator's opinion, make the subject inappropriate for this study
14. A person who is held in detention as the result of a judicial or official decision or who is in a subordinate relationship to the Sponsor or Investigator
15. A subject who, in the opinion of the Investigator, should not participate in the study for any reason, including if there is a question about the subject's ability to comply with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2021-09-16 (Actual); Primary Completion 2022-04-20 (Actual); Study Completion 2022-05-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dorothy Nguyen, MD, Study Chair — AmMax Bio, Inc.
Locations (5):
- AmMax Bio Clinical Site, Budapest, Hungary
- AmMax Bio Clinical Site, Warsaw, Poland
- Ukraine (3):
  - AmMax Bio Clinical Site, Dnipro
  - AmMax Bio Clinical Site, Kharkiv
  - AmMax Bio Clinical Site, Kyiv

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The original study design included multiple cohorts with an adaptive, dose escalation design. However, due to the early conclusion of the study, subjects were enrolled only in Cohort A, thus no additional dose cohorts were recruited.
Groups:
- Subjects With Tenosynovial Giant Cell Tumor: Cohort A: Received initial priming dose on Day 1 followed by 5 maintenance doses administered every 2 weeks (at Weeks 2, 4, 6, 8, and 10), for a total of 6 doses over the 12-week treatment period.
Period: Overall Study
Arm/Group | Subjects With Tenosynovial Giant Cell Tumor
Started | 4
Completed | 3
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: A total of 48 subjects were planned. However, enrollment into the study was stopped in November 2021 after 4 subjects were enrolled to focus more on AMB-05X intra-articular administration.
Groups:
- Cohort A: Subjects With TGCT: Low-Dose AMB-05X Each subject will receive a low dose of AMB-05X every 2 weeks, for a total of 6 doses over the 12-week treatment period.
  AMB-05X is a fully human antibody antagonist (immunoglobulin G, type 2 [IgG2]) specific to the extracellular domain of human CSF1R
Arm/Group | Cohort A: Subjects With TGCT
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Hungary | 1
  Ukraine | 2
  Poland | 1

OUTCOME MEASURES:

1. Primary Outcome: Treatment-emergent Adverse Events (TEAEs)
Description: The frequency and severity of reported TEAEs in Subjects with Tenosynovial Giant Cell Tumor (TGCT) receiving Intravenous AMB 05X.
Time Frame: 6 months
Population: All enrolled patients
Measure: Count of Participants; unit: Participants
Groups:
- Cohort A: Subjects With TGCT: AMB-05X Each subject will receive a 4mg/kg and maintenance dose of 2 mg/kg AMB-05X every 2 weeks, for a total of 6 doses over the 12-week treatment period.
  AMB-05X: A fully human monoclonal immunoglobulin (IgG2) directed against c-fms
Arm/Group | Cohort A: Subjects With TGCT
Number analyzed (Participants) | 4
Participants
  Number of subjects with treatment-emergent adverse events | 4
  Number of subjects without treatment-emergent adverse events | 0

2. Secondary Outcome: Overall Tumor Response (Objective Response) Per Response Evaluation Criteria in Solid Tumors (RECIST) v.1.1
Description: Response Evaluation Criteria in Solid Tumors (RECIST) v1.1; Per RECIST v1.0 for target lesions and assessed by MRI: A Complete Response (CR) is defined as disappearance of all tumors. A Partial Response (PR) is defined as at least a 30% decrease in the sum of diameters of target tumors from the baseline sum of diameters.
Time Frame: 12 weeks
Population: TGCT - Modified Intent-to-treat (ITT)- All TGCT subjects who received at least 1 dose of study drug and had both baseline and post-baseline data for at least 1 efficacy endpoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Subjects With TGCT
Number analyzed (Participants) | 3
Participants
  Subjects with CR | 0
  Subjects with PR | 1
  Subjects with stable disease | 2

3. Secondary Outcome: Overall Response Based on Tumor Volume Score (TVS)
Description: Tumor Volume Score (TVS) calculates tumor volume as a percentage of the estimated volume of the maximally distended synovial cavity or tendon sheath and provides a score in 10% increments. A score of 0 indicates no evidence of tumor; a score of 10 indicates a tumor that is equal in volume to that of a maximally distended synovial cavity or tendon sheath. Complete response (CR): lesion is completely gone; Partial response (PR): >/=50% decrease in TVS relative to Baseline; Progressive disease (PD): >/= 30% increase in TVS relative to the lowest score during the study; Stable disease (SD): does not meet any of the other classifications.
Time Frame: 24 weeks or ET visit
Population: TGCT - Modified Intent-to-treat (ITT) - All TGCT subjects who received at least 1 dose of study drug and had both baseline and post-baseline data for at least 1 efficacy endpoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Subjects With TGCT
Number analyzed (Participants) | 3
Participants
  Subjects with CR | 0
  Subjects with PR | 0
  Subjects with SD | 3

4. Secondary Outcome: Mean Change From Baseline Range of Motion (ROM) (Flexion, Knee) Scores
Description: Mean Change from Baseline in Range of Motion (ROM) Scores - Flexion (knee only). ROM is assessed by qualified assessors and recorded in degrees. At Baseline, the plane of movement with the smallest (worst) relative ROM was identified; only this plane was used for evaluating change in ROM. Higher scores indicate greater range of motion.
Time Frame: week 12
Population: Modified intent-to-treat, 3 subjects with ROM data in right and left knee were analyzed
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Subjects With TGCT
Number analyzed (Participants) | 3
Participants
  Subjects with no change in ROM from baseline | 1
  Subjects with change in ROM Left Knee | 1
  Subjects with change in ROM Right Knee | 1

5. Secondary Outcome: Mean Change From Baseline in the Patient-Reported Outcomes Measurement Information System (PROMIS) Physical Function Score
Description: Mean change from Baseline in the Patient-Reported Outcomes Measurement Information System (PROMIS) Physical Function score is used to assess physical function. PROMIS is a 10-question patient reported outcome instrument used to assess physical functioning based on use of the upper extremities (dexterity), lower extremities (walking or mobility), and central regions (neck, back) and on instrumental activities of daily living. Five questions address the degree to which the subject's health limits activities, and subjects select a response that ranges from 1-"cannot do" to 5-"not at all". Five additional questions address the degree to which the subject is able to perform certain physical activities, and subjects select a response to each question that ranges from 1 ("cannot do") to 5 ("without any difficulty"). Raw scores are summarized. The score range is 10 to 50, higher scores = worse physical function
Time Frame: 12 weeks
Population: Subjects with TGCT
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cohort A: Subjects With TGCT
Number analyzed (Participants) | 3
score on a scale | 0 (2.65)

6. Secondary Outcome: Serum Cmax for AMB-05X at Week 10 Post Dose
Description: The maximum concentration of AMB-05X in subject serum is measured at week 10 postdose, using sensitive enzyme-linked immunosorbent assay analyses (ELISA).
Time Frame: 10 weeks
Population: All enrolled subjects
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort A: Subjects With TGCT
Number analyzed (Participants) | 4
ng/mL | 54,457 (30,356)

7. Secondary Outcome: Number of Subjects With Anti-Drug Antibodies to AMB-05X at Week 10
Description: AMB-05X Anti-drug Antibodies (ADA) in subject serum will be measured from pre-dose samples.
Time Frame: 10 weeks
Population: All enrolled subjects
Measure: Count of Participants; unit: Participants
Arm/Group | Subjects With Tenosynovial Giant Cell Tumor
Number analyzed (Participants) | 4
Participants
  Subjects ADA positive at any visit analyzed | 1
  Subjects ADA negative at every visit analyzed | 3

8. Secondary Outcome: Mean Change From Baseline in Worst Stiffness Numeric Rating Scale (NRS) Score
Description: The mean changes from Baseline in the Worst Stiffness Numeric Rating Scale (NRS) score, a Patient-Reported Outcome (PRO) Measurement. The Worst Stiffness NRS is a single-item instrument designed to assess "worst" stiffness at the site of the tumor in the last 24 hours. The instrument uses an 11-point numeric rating scale that ranges from 0 ("no stiffness") to 10 ("stiffness as bad as you can imagine"). Higher scores indicate worse stiffness.
Time Frame: 12 weeks
Population: TGCT subjects
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cohort A: Subjects With TGCT
Number analyzed (Participants) | 3
score on a scale | -2.7 (2.52)

9. Secondary Outcome: Brief Pain Inventory Pain Severity Domain Score
Description: The mean changes from Baseline in Brief Pain Inventory (BPI) Pain Severity Domain. (Score of 0-10, where a negative score from baseline indicates a better BPI score, less severe pain) Brief Pain Inventory (BPI) is a self-administered questionnaire used to evaluate the severity of a subject's pain and the impact of this pain on the subject's daily functioning. For the Pain Severity domain the subject is asked to rate their worst, least, average, and current pain intensity, and list current treatments and their perceived effectiveness on a scale from 0 to 10, where higher scores mean more severe pain. All of the 0-10 scores are averaged to obtain the total Domain (subscale) Score.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cohort A: Subjects With TGCT
Number analyzed (Participants) | 3
score on a scale | -0.83 (1.665)

10. Secondary Outcome: Mean Change From Baseline in Brief Pain Inventory Severity Interference
Description: The mean changes from Baseline in Brief Pain Inventory (BPI) Severity Interference domain. The BPI Short Form is a patient-reported outcome instrument used to evaluate the severity of a subject's pain and the impact of this pain on the subject's daily functioning. For this domain, the subject is asked to rate their worst, least, average, and current pain intensity, list current treatments and their perceived effectiveness, and rate the degree that pain interferes with general activity, mood, walking ability, normal work, relations with other persons, sleep, and enjoyment of life on a scale from 0 to 10, where higher scores mean more pain interference. The reported score is the mean of the seven interference items. Higher scores indicate greater levels of pain.
Time Frame: 12 weeks
Population: TGCT subjects
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cohort A: Subjects With TGCT
Number analyzed (Participants) | 3
score on a scale | 0.81 (1.528)

11. Secondary Outcome: Worst Pain Numeric Rating Scale Score
Description: Mean change from Baseline in Worst Pain Numeric Rating Scale score. The Worst Pain Numeric Rating Scale is an item in the BPI that assesses a subject's "worst" pain in the last 24 hours. The 11-point Numeric Rating Scale for this item ranges from 0 ("no pain") to 10 ("pain as bad as you can imagine"). Higher scores indicate greater level of pain.
Time Frame: 12 weeks
Population: TGCT subjects
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cohort A: Subjects With TGCT
Number analyzed (Participants) | 3
score on a scale | -0.3 (1.53)

12. Secondary Outcome: EuroQol 5 Dimension 5 Level Health Assessment
Description: Mean change from Baseline in the EuroQol 5 Dimension 5 Level (EQ-5D-5L) assessment Scale Score (5-25). This instrument is a self-report survey that measures quality of life across 5 domains: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension is scored on a 5-level severity ranking that ranges from "no problems" through "extreme problems". Higher scores indicate a lower quality of life.
Time Frame: 12 weeks
Population: TGCT subjects
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cohort A: Subjects With TGCT
Number analyzed (Participants) | 3
score on a scale | -0.3 (0.58)

13. Secondary Outcome: Colony-stimulating Factor 1 Levels
Description: Serum colony-stimulating factor-1 (CSF-1) levels are measured in patient/subject serum. Samples were collected for measurement of CSF-1 at least once at specified visits.
Time Frame: 10 weeks
Population: TGCT subjects
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Cohort A: Subjects With TGCT
Number analyzed (Participants) | 3
pg/mL | 1216 (372)

14. Secondary Outcome: Mean Change From Baseline Rnge of Motion (Flexion, Ankle) Scores
Description: Mean Change from Baseline in Range of Motion (ROM) Scores - Flexion (Ankle only). ROM is assessed by qualified assessors and recorded in degrees. At Baseline, the plane of movement with the smallest (worst) relative ROM was to be identified; only this plane was used for evaluating change in ROM. Higher scores indicate greater range of motion.
Time Frame: week 12
Population: Although the protocol allowed patients with TGCT of the ankle, no subjects with TGCT of the ankle were enrolled.
Arm/Group | Subjects With Tenosynovial Giant Cell Tumor
Number analyzed (Participants) | 0

15. Secondary Outcome: Serum AMB-05X-Binding Anti-drug Antibody (ADA) Levels
Description: Series analysis for anti-drug antibody detection and titer
Time Frame: Week 12
Population: Measurement of serum AMB-05X-Binding anti-drug antibody (ADA) levels was a prespecified secondary outcome measure. ADA data for 4 subjects enrolled prior to study termination are provided. One of 4 subjects provided only a baseline sample. Three of 4 subjects provided both baseline (Visit 2) and Week 10 (Visit 7) samples. No conclusions were made based on the limited information collected at study termination (Sponsor stopped developing intravenous AMB-05X for patients with TGCT).
Measure: Count of Participants; unit: Participants
Arm/Group | Subjects With Tenosynovial Giant Cell Tumor
Number analyzed (Participants) | 4
Participants
  Baseline visit: Subjects ADA negative | 3
  Baseline visit: Subjects ADA positive | 1
  Visit 7: number analyzed (Participants) | 3
  Visit 7: Subjects ADA negative | 2
  Visit 7: Subjects ADA positive | 1

ADVERSE EVENTS:
Time Frame: 6 months
Groups:
- Tenosynovial Giant Cell Tumor - Events During Initial Treatment Period; Tenosynovial Giant Cell Tumor - Events During Maintenance Treatment Period: Cohort A: Received initial priming dose on Day 1 followed by 5 maintenance doses administered every 2 weeks (at Weeks 2, 4, 6, 8, and 10), for a total of 6 doses over the 12-week treatment period.
Arm/Group | Tenosynovial Giant Cell Tumor - Events During Initial Treatment Period | Tenosynovial Giant Cell Tumor - Events During Maintenance Treatment Period
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 0/4 | 4/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tenosynovial Giant Cell Tumor - Events During Initial Treatment Period (N=4) | Tenosynovial Giant Cell Tumor - Events During Maintenance Treatment Period (N=4)
face edema (General disorders) | 0 (0) | 4 — Face Edema
hepatic enzyme increased (Investigations) | 0 | 1 — elevated liver enzymes
epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
hypertension (Vascular disorders) | 0 | 1
headache (Nervous system disorders) | 0 | 1
rash maculopapular (Skin and subcutaneous tissue disorders) | 0 | 1
skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 1
blood lactate dehydrogenase increased (Investigations) | 0 | 2
diarrhea (Gastrointestinal disorders) | 0 | 1
aspartate aminotransferase increased (Investigations) | 0 | 1
pyelonephritis acute (Infections and infestations) | 0 | 1
urinary tract infection (Infections and infestations) | 0 | 1

LIMITATIONS AND CAVEATS:
A decision was made in November 2021 to stop further enrollment into the study to allow development to focus on AMB-05X intra-articular administration for TGCT. A total of 4 subjects had been enrolled into the study at the time the decision to cease further enrollment was made, limiting the ability to interpret the resulting data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-18): https://cdn.clinicaltrials.gov/large-docs/80/NCT04938180/Prot_SAP_001.pdf